CLINICAL TRIAL: NCT05364502
Title: A Prospective Multicenter Single-Arm Staged Study to Evaluate the Safety and Effectiveness of Embrace™ Hydrogel Embolic For Transcatheter Embolization of Arterial Bleeding in Solid Organs and Peripheral Arteries
Brief Title: (HALT) Embrace Hydrogel Embolic System (HES) Study of Embolization in Peripheral Arterial Bleeds
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instylla, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INY-P-21-002
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-07

CONDITIONS: Arterial Bleeding in Solid Organs and Peripheral Arteries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Embrace HES including Instylla™ Delivery Kit and Instylla™ Microcatheter — The Embrace Hydrogel Embolic System (HES) is indicated for embolization of peripheral arterial bleeds in vessels ≤6mm

SUMMARY:
To evaluate the safety and effectiveness of Embrace Hydrogel Embolic System for the transcatheter embolization of peripheral arterial bleeds.

DETAILED DESCRIPTION:
A Prospective Multicenter Single-Arm Staged Study to Evaluate the Safety and Effectiveness of Embrace™ Hydrogel Embolic For Transcatheter Embolization of Arterial Bleeding in Solid Organs and Peripheral Arteries

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age ≥ 18 years old
2. Subjects who are candidates for transarterial catheter embolization with arterial bleeding documented on a suitable radiologic imaging and/or endoscopic visualization study taken during the index hospitalization that allows for the source of the arterial injury/bleeding to be localized. Includes (but not limited to) the following:

   1. Non-variceal Upper Gastrointestinal (UGI) bleeds refractory to endoscopic treatment
   2. End organ/visceral bleeds (kidney, liver and spleen including tumor bleeds)
   3. Spontaneous hematoma (e.g., rectus sheath and psoas muscle hematomas)
   4. Other peripheral arterial bleeds (e.g., pelvic hemorrhage) if not associated with risk of ischemia distal to the lesion or embolization of non-expendable arteries.
3. Subjects with at least one target vessel ≤6mm and Embrace HES can be delivered to the target vessel(s).
4. Subject is willing to comply with follow-up evaluation schedule.
5. No prior embolization in the target territory prior to study entry
6. The subject or a legally authorized representative has provided informed consent approved by the appropriate local IRB/EC.

Exclusion Criteria:

1. Life expectancy ≤ 30 days
2. In the Investigator's opinion, due to injury severity the subject is not likely to benefit from angioembolization (e.g., in the presence of significant polytrauma, multiple organ failure or shattered organs).
3. Any contraindication to arteriography or the embolization protocol utilized at treating institution.
4. Pregnant or breast-feeding (women of child-bearing potential must undergo a pregnancy test performed in accordance with local institutional requirements and agree to use contraception for at least six months).
5. Hemorrhagic shock (Class IV-see Appendix 1) at time of treatment
6. Target vascular territory supplied by the pulmonary artery, coronary artery, or cerebral or cerebellar artery (requiring embolization of these arteries) or the artery to be embolized has connections to these arteries via a collateral pathway.
7. Embolization for treatment of spinal arteries, lower GI bleeds, arteriovenous malformations, embolization of arteriovenous shunts, endoleak management, neurovascular bleeds, penetrating trauma of extremities.
8. Forrest Classification Type III UGI bleeds (see Appendix 2)
9. In the investigator's opinion, patient will require embolization of 4 or more discrete vascular territories/arterial injuries (requires that microcatheter be repositioned to discrete area) based on diagnostic angiography or another suitable imaging study.
10. Known or suspected angio-anatomical conditions that in the Investigator's opinion, would prevent the delivery catheter to gain access to the selected position for safe and intended embolization.
11. Known allergies (based on history) to PEG, ferrous compounds, tert Butyl Hydroperoxide, contrast media or procedural sedatives/anesthetics that is not amenable to pre-medication
12. Presence of medically relevant localized or systemic infection
13. The patient has other concurrent conditions or known history that in the opinion of the Investigator would be unlikely to receive clinical benefit from the study procedure or participation in the study may compromise patient safety or study objectives (including but not limited to ongoing acute infection, life-threatening concomitant trauma or conditions).
14. Presence of Uncorrectable Coagulopathy: Defined as thrombocytopenia with platelet counts < 40,000/mm3 and/or INR > 2.0.
15. If known, enrollment in a concurrent study in which the study treatment may confound the evaluation of the study device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint | Through 30 days post-index procedure
  Freedom from major adverse events (MAE)
Clinical Success | Within 30 days of the index procedure
  Defined as the absence of bleeding from the target lesion after embolization with Embrace HES without the need for subsequent embolic devices in the index procedure, emergency surgery, re-embolization or other target vessel re-interventions due to rebleeding.
Technical Success | Immediately following index procedure
  Defined as occlusion of the target vessel or exclusion of the area of arterial damage and/or the cessation of extravasation on angiography after embolization with Embrace HES.

CONTACTS AND LOCATIONS:
Overall Officials: Suvranu Ganguli, Principal Investigator — Boston Medical Center
Locations (22):
- United States (22):
  - Banner Health, Phoenix, Arizona
  - Memorial Health Services, Long Beach, California
  - Stanford University, Stanford, California
  - UCLA Harbor Lindquist Institute, Torrance, California
  - Nuvance Health, Danbury, Connecticut
  - Yale University, New Haven, Connecticut
  - Medstar Georgetown University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Northwestern, Evanston, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Mount Sinai Hospital, New York, New York
  - Columbia University Milstein, New York, New York
  - UNC School of Medicine, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Medical College of Wisconsin, Milwaukee, Wisconsin